CLINICAL TRIAL: NCT00442793
Title: A Randomized, Open Label Study Comparing the Effect of Mircera and Epoetin Beta on Hemoglobin Response in Patients With Chronic Kidney Disease Who Are on Dialysis
Brief Title: A Study Comparing Mircera and Epoetin Beta for the Treatment of Anemia in Dialysis Patients With Chronic Kidney Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20680
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta; continuous erythropoietin receptor activator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: Epoetin beta

INTERVENTIONS:
Drug: Epoetin beta — As prescribed, 3 times weekly
  Arms: 2
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 0.4 micrograms/kg iv every 2 weeks
  Arms: 1

SUMMARY:
This 2 arm study will compare the effect on hemoglobin response of Mircera and epoetin beta, in patients with chronic renal anemia who are on dialysis. Eligible patients will be randomized to receive either Mircera (0.4 micrograms/kg i.v. every 2 weeks) or epoetin beta (3 times weekly, according to approved labelling). The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia requiring dialysis;
* maintenance hemodialysis or peritoneal dialysis for >=2 weeks before and during screening;
* adequate iron status.

Exclusion Criteria:

* previous epoetin treatment within 8 weeks prior to screening;
* failing renal graft in place;
* bleeding episode necessitating transfusion within 8 weeks prior to screening;
* poorly controlled hypertension;
* previous treatment with Mircera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Hb response rate | Weeks 0-24
Change in Hb concentration between baseline and evaluation period | Months 4-6

SECONDARY OUTCOMES:
Hb over time | Throughout study
Time to Hb response | Throughout study
RBC transfusions | Weeks 0-24
AEs, laboratory parameters, vital signs | Throughout study
Serum concentration of Mircera | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (6):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
- Hong Kong, Hong Kong